CLINICAL TRIAL: NCT02034097
Title: A Phase II Study to Evaluate Foretinib in Genomic Subpopulations of Subjects With Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: A Study to Evaluate Foretinib in Subjects With Non-Small-Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: GSK has decided to terminate the Product Development of foretinib and conclude our Development Agreement with Exelixis
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112132
Record Dates: First submitted 2013-11-27; First posted 2014-01-13 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Cancer
Keywords: ROS1; erlotinib; EGFR; non-small cell lung cancer; foretinib
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — GSK 1363089; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Subjects with EGFRm NSCLC who have received clinical benefit (CR, PR, SD) for at least 4 months and then progressed on an EGFR-TKI within the last 30 days will receive 150 milligram (mg) erlotinib once daily (OD) and 45 mg foretinib OD as a combination therapy until disease progression
  Interventions: Drug: Foretinib; Drug: Erlotinib
- Cohort 2 (Experimental): Subjects with EGFR/WT NSCLC who have received clinical benefit (CR, PR, SD) for at least 2 months and then progressed on an EGFR-TKI within the last 30 days will receive 150 mg erlotinib OD and 45 mg foretinib OD as a combination therapy until disease progression.
  Interventions: Drug: Foretinib; Drug: Erlotinib
- Cohort 3 (Experimental): Subjects with NSCLC who are predicted to be sensitive to foretinib based on biomarkers identified with preclinical or clinical data will receive 60 mg foretinib OD as a monotherapy until disease progression
  Interventions: Drug: Foretinib

INTERVENTIONS:
Drug: Foretinib — Round yellow tablet containing 15 mg of foretinib will be orally administered in a dose level of 45 mg (3 x 15 mg) or 60 mg (4 x 15 mg) OD until disease progression
Drug: Erlotinib — Round white tablet containing either 25 mg, 100 mg, or 150 mg of erlotinib will be orally administered in a dose level of 150 mg OD until disease progression
  Arms: Cohort 1; Cohort 2

SUMMARY:
Foretinib (GSK1363089) is an investigational, oral, multikinase inhibitor involved in invasion, migration, and angiogenesis. This is a phase II, open label, uncontrolled, parallel, multi-cohort, multicenter 2-stage study to assess the safety and efficacy of foretinib and erlotinib combination therapy and foretinib monotherapy in genomic subpopulations of Non-Small-Cell Lung Cancer (NSCLC) subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent, approved by the Independent Ethics Committee (IEC) or Institutional Review Board (IRB), obtained prior to the performance of any study-specific procedures or assessments. The subject must be able to understand and comply with protocol requirements and instructions.
* Males and females >=18 years of age (at the time consent is obtained).
* Histologically or cytologically documented stage IV NSCLC, with prior histopathological reports showing one of the following: Evidence of Epidermal growth factor receptor activating mutation positive (EGFRm) or Epidermal growth factor receptor (EGFR)/ Wild Type (WT) genes in Deoxyribonucleic acid (DNA) derived from formalin-fixed paraffin-embedded human non-small cell lung cancer tumor tissue; An orphan receptor tyrosine kinase (ROS1) chromosomal rearrangements as determined by ectopic expression of the ROS1 protein by immunohistochemistry (IHC) and/or detection of ROS1 rearrangements as determined by Fluorescence in situ hybridization (FISH); In Cohort 3, subjects with alternative molecular profiles (e.g., Non-receptor tyrosine kinases [NRTK], Tyrosine kinase receptor for members of the glial cell line-derived neurotrophic factor (GDNF) family [RET], etc.) may be enrolled as subsets of this cohort if emerging data suggest they would likely respond to therapy. If genetic analyses have been performed previously, a copy of the complete mutation profile is requested.
* Tumor biopsy: For Cohort 1 and Cohort 2, a fresh tumor sample after progression on erlotinib, gefitinib, afatinib, or another EGFR- Tyrosine kinase inhibitors (TKI) and before starting in this study is required; in addition, archival samples obtained pre-EGFR-TKI are required (if available). For Cohort 3, subjects who are crizotinib/ROS1 inhibitor naive will be required to provide a copy of the genetic report showing ROS1 positive mutation and archival tissue if available; subjects with ROS1 fusions who progressed on crizotinib/ROS1 inhibitor will be required to provide a copy of the genetic report showing ROS1 positive mutation and a fresh biopsy.
* Subjects must meet one of the following: Cohort 1 (EGFRm): Has documented progression (based on RECIST 1.1 criteria) after >=4 months of clinical benefit on prior erlotinib/gefitinib/afatinib therapy within 30 days prior to the first dose of foretinib; Cohort 2 (EGFR/WT): Has documented progression (based on RECIST 1.1criteria) after >=2 months of clinical benefit on prior EGFR-TKI therapy within 30 days prior to the first dose of foretinib, or; Cohort 3: For the ROS1 subset, documented progression (based on RECIST 1.1 criteria) on or was intolerant of prior crizotinib/ROS1 inhibitor therapy or is naive to crizotinib/ROS1 inhibitor. Note: Crizotinib/ROS1 inhibitor naive subjects will be eligible for the study if crizotinib/ROS1 inhibitor is not available to them and participation in this trial is their only option for targeted ROS1 treatment. For additional biomarker-driven subsets, written documentation of entry requirements will be provided to IRB(s)/IEC(s).
* Only one prior line of EGFR-TKI therapy immediately preceding enrolment into the current study for Cohorts 1 or 2. Progression will have occurred on single agent EGFR-TKI treatment in the 1st line setting for EGFRm subjects, and in the 2nd line or maintenance setting for EGFRm or EGFR/WT subjects.
* Measurable disease, i.e., presenting with at least one measurable lesion per RECIST v1.1.
* Subjects must not have participated in another clinical trial except with single agent EGFR-TKI or crizotinib/ROS1 inhibitor within the past 3 months and may not have received any intervening therapy of any kind (chemotherapy, immunotherapy, etc.) between the time of progression on prior TKI and enrolment on this trial. Additional requirements regarding prior therapy may be added for Cohort 3 subsets as they are added to this study. Note: Subjects may continue treatment with the prior TKI on which they progressed during this 30 day period at the discretion of investigator, but must discontinue the prior TKI to allow 5 half-lives off drug prior to the first dose of foretinib in this study.
* A minimum of 14 days must have elapsed since any palliative radiotherapy and subjects must have recovered from any treatment related toxicities prior to enrolment.
* A minimum of 14 days has elapsed from last surgery prior to first dose and wound healing has occurred. If subject has had exploratory thoracotomy, they must have recovered from the procedure prior to start.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Any ongoing potentially reversible treatment-related toxicities must be (National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03) <=Grade 1 and not progressing in severity, except alopecia or the expected EGFR-TKI toxicities of rash or diarrhea that are stable with intervention and then only if agreed to by the GlaxoSmithKline (GSK) Medical Monitor and the investigator.
* Adequate baseline organ function as defined in the protocol. Note: Laboratory results obtained during Screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the investigator may opt to retest the subject and the subsequent within range screening result may be used to confirm eligibility.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception, as defined in the protocol, during the study and for 21 days following the last dose of study treatment.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception as described in the protocol for at least 14 days prior to administration of the first dose of study until 21 days after the last dose of study treatment to allow for clearance of any altered sperm.
* Subjects must discontinue hormone replacement therapy prior to study enrolment due to the potential for inhibition of cytochrome P450 enzymes that metabolize estrogens and progestins.
* Cotinine level within the quantification limits of the assay. Subjects in erlotinib combination cohorts must have stopped smoking prior to study entry and must not have used any nicotine-containing products, including nicotine patches or gum, within the past 6 months.
* Able to swallow and retain orally administered study treatment.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Lactating female.
* Active malignancies other than the disease under study within the past 3 years, except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
* Subjects with untreated brain or meningeal metastases are not eligible (computerized tomography [CT] scans are not required to rule this out unless there is a clinical suspicion of central nervous system [CNS] disease). Subjects with treated and radiologic or clinical evidence of stable brain metastases (confirmed by 2 scans at least 4 weeks apart), with no evidence of cavitation or hemorrhage in the brain lesion are eligible providing that they are asymptomatic and do not require corticosteroids.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent, or compliance to the study procedures, in the opinion of the investigator or GSK Medical Monitor.
* Current use of a prohibited medication or requirement for any of these medications during treatment with foretinib or erlotinib.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to foretinib or erlotinib or excipients that in the opinion of the investigator or GSK Medical Monitor contraindicate their participation.
* Presence of active gastrointestinal disease (including Gastrointestinal [GI] bleeding or ulceration) or other condition that could affect GI absorption (e.g., malabsorption syndrome), history of biliary tract disease, or presence of uncontrolled emesis.
* Evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
* Subjects with appreciable cavitation in central thoracic lesions or lesion abutting a major blood vessel are not eligible. Subjects with overt bleeding from any site (>30 milliliter [mL] bleeding/episode) within 3 months of study entry are not eligible. No clinically relevant hemoptysis (>5 mL fresh blood) within 4 weeks prior to study entry is permitted. Subjects with only flecks of blood in sputum are permitted. Any questions about these criteria should be directed to the GSK Medical Monitor prior to registration.
* Corrected QT interval (QTc) >=470 milliseconds (msecs). Other clinically significant ECG abnormalities including 2nd degree (type II) or 3rd degree atrioventricular (AV) block.
* History of pulmonary embolism (PE) or deep venous thrombosis (e.g., calf vein thrombosis) within the past 6 months except subjects with recent Deep vein thrombosis (DVT) who have been treated with therapeutic anticoagulating agents for at least 6 weeks. If medically appropriate and treatment available, the investigator should consider switching these subjects to low molecular weight (LMW) heparin.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within the past 6 months.
* Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system. Subjects who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Subjects with a significant cardiac history (even if controlled) or prior doxorubicin exposure are required to have a Left Ventricular Ejection Fraction (LVEF) >=50%.
* Subjects with resting blood pressure (BP) consistently higher than systolic >140 millimeters of mercury (mmHg) and/or diastolic >90 mmHg (in the presence or absence of a stable dose of antihypertensive medication) or poorly controlled hypertension, history of labile hypertension or poor compliance with anti-hypertensive medication.
* French subjects: The French subject has participated in any study using an investigational study treatment(s) during the previous 30 days.
* Consumption of Seville oranges, grapefruit or grapefruit juice, and pomelos from 7 days prior to the first dose of study treatment(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Screening, Cycle 3 Day 1, Cycle 5 Day 1, then every 3 cycles up to 2 years
  ORR (confirmed Complete Response [CR] or confirmed partial response [PR]) will be assessed by investigator as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

SECONDARY OUTCOMES:
Number of subjects with adverse events | From the first dose of study treatment up to 2 years
Clinical laboratory tests | From screening up to 2 years
  Clinical laboratory assessments will include haematology, clinical chemistry and urinalysis parameters
Physical examinations | From screening up to 2 years
  Physical examinations will include assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities
Vital signs | From screening up to 2 years
  Vital sign measurements will include systolic and diastolic blood pressure and pulse rate
12-lead electrocardiograms (ECGs) | From screening up to 2 years
  Single 12-lead ECGs will be obtained at the scheduled time points
Electroretinogram (ERG) assessments | From screening up to 2 years
  A thorough eye examination, including electroretinogram will be performed at the scheduled time points
Clinical benefit rate | Screening, Cycle 3 Day 1, Cycle 5 Day 1, then every 3 cycles up to 2 years
  Clinical benefit rate is the percentage of subjects with CR + PR + stable disease (SD)
Length of clinical benefit, Length of SD, Length of progression-free survival (PFS), length of survival from first dose to death | Screening, Cycle 3 Day 1, Cycle 5 Day 1, then every 3 cycles up to 2 years
Population pharmacokinetic (PK) parameters | Cycle 1 Day 8 and Cycle 1 Day 15
  Population PK parameters including the apparent clearance following oral dosing (CL/F), apparent volume of distribution following dosing (Vd/F), and the effect of combination therapy on CL/F will be estimated

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline